CLINICAL TRIAL: NCT04034329
Title: PREservation Versus Thermal Ablation of the Incompetent Great Saphenous Vein in Varicose Veins Treatment
Brief Title: PREservation Versus Thermal Ablation
Acronym: PRETA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Ihar Ihnatovich, Professor, Belarusian State Medical University
Other Study IDs: 20140451
Record Dates: First submitted 2019-07-23; First posted 2019-07-26 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Varicose Veins
Keywords: ASVAL; EVLA; GSV; Long-term efficacy
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASVAL - group: GSV diameter ≤ 6 mm
  Interventions: Procedure: ASVAL
- EVLA-group: GSV diameter > 6 mm
  Interventions: Procedure: EVLA

INTERVENTIONS:
Procedure: ASVAL — Ambulatory Selective Varices Ablation under Local Anesthesia
  Groups: ASVAL - group
Procedure: EVLA — Endovenous Laser Ablation
  Groups: EVLA-group

SUMMARY:
This study will be looking at the effect of Ambulatory Selective Varices Ablation under Local Anesthesia (ASVAL) and Endovenous Laser Ablation (EVLA) with concomitant phlebectomy in patients with incompetent great saphenous vein (GSV).

DETAILED DESCRIPTION:
Full venous duplex ultrasonography was performed using Medical ultrasound scan. Cognizant of the negative consequences of standing and sitting for long periods of time (e.g. venous hypertension, venous reflux), we scheduled investigations for early morning, thus ensuring examination of the physiological status of the venous system in each patient. Ultrasound examinations of reflux at the saphenofemoral junction (SFJ) were performed using the Valsalva maneuver. Ultrasound examination of GSV reflux was performed by manually compressing the calf followed by sudden release. Reverse flow that lasted more than 0.5 seconds was considered pathological. Preoperative venous duplex mapping was done in the upright position. Further measurements of the GSV diameter 15 cm below the SFJ level were conducted to describe the severity of varicose veins more accurately.

The diameter of GSV at the 15-cm below the SFJ level was the main criterion to identify two groups of patients. Those with the GSV diameter ≤ 6 mm were treated with ASVAL. If the diameter of GSV was > 6 mm, EVLA with concomitant phlebectomy was performed.

All surgical procedures were accomplished by the same surgeon, using tumescent local anesthesia (i.e. 0,1% lidocaine and sodium bicarbonate solution without epinephrine).The EVLA was done under duplex guidance with a 1560-nm diode laser using bare fibres via a Seldinger wire technique. The GSV was cannulated at the lowest point of the reflux. The laser fiber was advanced below the SFJ at the level of v. epigastrica sup. after which the GSV was ablated during gradual withdrawal of the fibre. The 15 Watts laser power was delivered in a continuous pull back traction. The average applied linear endovenous energy dose (LEED) was 75,3 J/cm.

Peripheral side branches were removed by multiple stab avulsions in both groups. After the treatment, the leg was wrapped in sterile absorbent bandages, and compression stockings class II (23-32 mm Hg) were put on and recommended to wear for two weeks. All patients were discharged on the day of the treatment and were invited to a follow-up duplex ultrasonography (DUS) on the 1st post-operative day, 2 years and 5 years after the operation (patients were contacted by phone). DUS at follow-up visits was carried out by an independent specialist who was not involved in the initial treatment of the patients. To report clinical recurrence after EVLA we have used Group d' Evaluation des Lasers et de l'Echographie Vasculare (GELEV) score.

ELIGIBILITY:
Inclusion Criteria:

* Great saphenous vein (GSV) incompetence with reflux at least down to the knee level
* Primary symptomatic varicose veins, Clinical Etiological Anatomical Pathophysiological (CEAP) classification, clinical class C2-C3
* Physical status according to American Society of Anesthesiologists (ASA) I-II (I-Healthy, non-smoking, no or minimal alcohol use; II-Mild diseases only without substantive functional limitations)

Exclusion Criteria:

* Previous surgical groin exploration, except herniotomy
* Small saphenous vein, anterior or posterior accessory saphenous vein incompetence at the same limb
* Deep venous thrombosis, thrombophilia associated with a high risk of deep venous thrombosis or postthrombotic syndrome
* Arterial occlusive disease more severe than Intermittent claudication after more than 200 meters of pain free walking (Fontaine IIA) and/or ankle brachial index below 0.8

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GSV incompetence and C2-C3 were included in the prospective consecutive case study if they satisfied the selection criteria
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with pain or other discomfort (ie aching, heaviness, fatigue, soreness, burning) from absent (score 0) to severe (score 3) | 2-5 years
  None (0), Occasional (1), Daily, interfering with, but not preventing regular daily activities (2), Daily limiting most regular daily activities (3)
Number of Participants with varicose Veins from absent (score 0) to severe (score 3). | 2-5 years
  None (0), Few, scattered (1), Confined to calf or thigh (2) Involve calf and thigh (3)
Number of Participants with venous oedema from absent (score 0) to severe (score 3). | 2-5 years
  None (0) Limited to foot or ankle (1), Extends above ankle but below knee (2), Extends to knee or above (3)
Number of Participants with skin Pigmentation from absent (score 0) to severe (score 3). | 2-5 years
  None (0), Limited to perimalleolar area (1), Diffuse over lower third of calf (2), Wider distribution (above lower third of calf) (3)
Number of Participants with inflammation from absent (score 0) to severe (score 3). | 2-5 years
  None (0), Limited to perimalleolar area (1), Diffuse over lower third of calf (2), Wider distribution (above lower third of calf) (3)
Number of Participants with induration from absent (score 0) to severe (score 3). | 2-5 years
  None (0), Limited to perimalleolar area (1), Involving lower third of calf (2), Involving more than lower third of calf (3)
Number of Participants with active ulcers from absent (score 0) to severe (score 3). | 2-5 years
  None (0), 1 (1), 2 (2), more than 2 (3)
Number of Participants with different duration of active ulcer: from absent (score 0) to severe (score 3). | 2-5 years
  None (0), Less than 3 months (1), More than 3 months but less than 1 year (2) More than 1year (3)
Number of Participants with active ulcer diameter from absent (score 0) to severe (score 3). | 2-5 years
  None (0), Diameter less than 2 cm (1), Diameter 2-6 cm (2), Diameter more than 6 cm (3)
Number of Participants with compression therapy from absent (score 0) to severe (score 3). | 2-5 years
  Not used (0), Intermittent use of stockings (1), Uses stockings most days (2), Full compliance with stockings (3)

SECONDARY OUTCOMES:
Number of Participants with clinical recurrence-free rate (no - score 0, yes - score 1) | 2-5 years
  Visible or palpable varicosity with a diameter of less than 3 mm after surgery (0). Visible or palpable varicosity with a diameter of more than 3 mm after surgery (1).

CONTACTS AND LOCATIONS:
Overall Officials: Genadz Kandratsenka, Prof, Study Chair — Educational Institution"Belarusian State Medical University"
Locations (1):
- Educational Institution"Belarusian State Medical University", Minsk, Dzerzhinski Ave., 83, Belarus

IPD SHARING:
Plan to Share IPD: Yes
To compare clinical efficacy of Ambulatory Selective Varices Ablation under Local Anesthesia (ASVAL) and Endovenous Laser Ablation (EVLA) with concomitant phlebectomy in patients with incompetent great saphenous vein (GSV).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 01.2020
Access Criteria: To compare clinical efficacy of Ambulatory Selective Varices Ablation under Local Anesthesia (ASVAL) and Endovenous Laser Ablation (EVLA) with concomitant phlebectomy in patients with incompetent great saphenous vein (GSV).

REFERENCES:
- [Background] Pittaluga P, Chastanet S. Persistent incompetent truncal veins should not be treated immediately. Phlebology. 2015 Mar;30(1 Suppl):98-106. doi: 10.1177/0268355515569141. PMID 25729076
- [Background] Chastanet S, Pittaluga P. Influence of the competence of the sapheno-femoral junction on the mode of treatment of varicose veins by surgery. Phlebology. 2014 May;29(1 suppl):61-65. doi: 10.1177/0268355514529207. Epub 2014 May 19. PMID 24843088
- [Background] van Neer P, Kessels FG, Estourgie RJ, de Haan EF, Neumann MA, Veraart JC. Persistent reflux below the knee after stripping of the great saphenous vein. J Vasc Surg. 2009 Oct;50(4):831-4. doi: 10.1016/j.jvs.2009.05.021. Epub 2009 Jul 12. PMID 19595549
- [Background] Zolotukhin IA, Seliverstov EI, Zakharova EA, Kirienko AI. Short-term results of isolated phlebectomy with preservation of incompetent great saphenous vein (ASVAL procedure) in primary varicose veins disease. Phlebology. 2017 Oct;32(9):601-607. doi: 10.1177/0268355516674415. Epub 2016 Oct 19. PMID 27760806
- [Background] Harlander-Locke M, Jimenez JC, Lawrence PF, Derubertis BG, Rigberg DA, Gelabert HA. Endovenous ablation with concomitant phlebectomy is a safe and effective method of treatment for symptomatic patients with axial reflux and large incompetent tributaries. J Vasc Surg. 2013 Jul;58(1):166-72. doi: 10.1016/j.jvs.2012.12.054. Epub 2013 Apr 6. PMID 23571079
- [Background] Puggioni A, Kalra M, Carmo M, Mozes G, Gloviczki P. Endovenous laser therapy and radiofrequency ablation of the great saphenous vein: analysis of early efficacy and complications. J Vasc Surg. 2005 Sep;42(3):488-93. doi: 10.1016/j.jvs.2005.05.014. PMID 16171593
- [Background] Nesbitt C, Bedenis R, Bhattacharya V, Stansby G. Endovenous ablation (radiofrequency and laser) and foam sclerotherapy versus open surgery for great saphenous vein varices. Cochrane Database Syst Rev. 2014 Jul 30;(7):CD005624. doi: 10.1002/14651858.CD005624.pub3. PMID 25075589